CLINICAL TRIAL: NCT00044720
Title: An Open-label, Concentration Controlled, Randomized, 12 Month Study of Prograf + Rapamune + Cor
Brief Title: Study Evaluating Sirolimus in End Stage Renal Disease in High Risk Kidney Transplant Recipients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Masking: None
Other Study IDs: 0468H1-101164
Record Dates: First submitted 2002-09-04; First posted 2002-09-06 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Kidney Failure; Graft vs Host Disease; Kidney Transplantation
Keywords: Kidney Transplant
MeSH Terms: conditions — Kidney Failure, Chronic; Graft vs Host Disease | interventions — Sirolimus

INTERVENTIONS:
Drug: Rapamune

SUMMARY:
The incidence of efficacy failure at 12 months between two regimens.

ELIGIBILITY:
Inclusion Criteria

* Age: 13 years or older, 40 kgs or more
* End-stage renal disease
* African-American/Black transplant recipient and/or repeat renal transplant recipient who lost a previous allograft

Exclusion Criteria

* Evidence of active infection
* Evidence abnormal chest x-ray
* Patients with HIV.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 484 (Actual)
Dates: Primary Completion 2005-07 (Actual); Study Completion 2005-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, MD, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer